CLINICAL TRIAL: NCT03572920
Title: Actigraphy-based RAR and Sleep Behavior in Hospitalized Patients for Hip/Knee Prosthesis
Brief Title: Sleep Behavior and Rest-activity Circadian Rhythm (RAR) in Hip/Knee Prosthesis
Acronym: Sleep&RAR
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Sonno&protesi
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2018-07

CONDITIONS: Sleep; Pain; Hospitalization; Arthroplasty Complications; RAR
Keywords: Sleep; Actigraphy; Pain; Patients; Hospitalization; Hip Replacement; Knee Replacement; Arthroplasty; RAR
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hip/knee arthroplasty.: RAR description by actgraphy Objective sleep evaluation by actigraphy. Subjective sleep quality with sleep diary Pittsburgh Sleep Quality Index (PSQI).
  Interventions: Device: Objective sleep evaluation by actigraphy; Other: Pittsburgh Sleep Quality Index (PSQI)

INTERVENTIONS:
Device: Objective sleep evaluation by actigraphy — Each subject will wear a wrist activity monitor (actigraphy) to detect his/her sleep behaviour during hospitalization.
Other: Pittsburgh Sleep Quality Index (PSQI) — Each subject will fill twice the Pittsburgh Sleep Quality Index (PSQI), before hospitalization and after the 10th day, to evaluate his/her subjective sleep quality.

SUMMARY:
The consequences of chronically insufficient sleep are both behavioral and medical. . Patients who undergo total knee or hip arthroplasty commonly complain of sleep fragmentation after hospitalization The aim of the present study is to evaluate the changes inrest-activity circadian rhythm (RAR) and objective and subjective sleep quality and perceived pain, untill the 10th hospitalization day, in patients who underwent total knee or hip arthroplasty.

DETAILED DESCRIPTION:
The National Health and Nutrition Examination Survey found that 22% of the US population reported 6 h of sleep or less and another 15% registered 5 h of sleep or less per 24 h (1). The consequences of chronically insufficient sleep are both behavioral and medical. Quantity and quality of sleep represent important factors for the quality of life, which can have positive or negative influence on individual health (2-4). Patients who undergo total knee or hip arthroplasty commonly complain of sleep fragmentation after hospitalization (5,6) Such patients experience acute postsurgical pain and discomfort, including restriction of their leg movement to prevent dislocation of the hip implant in the acute stage. The results of previous post-surgery studies have shown that REM sleep was severely reduced and awake time increased on the first postoperative night compared with the preoperative night (7,8).It is necessary for patients to secure the appropriate amount and quality of sleep to facilitate recuperation after surgery. Sleep disturbance is also related to the presence of delirium. The aim of the present study is to evaluate the changes in objective and subjective sleep quality and perceived pain, untill the 10th hospitalization day, in patients who underwent total knee or hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Male of female subjects aged between 50 and 80 years old.
* Knee or Hip Arthroplasty at IRCCS Galeazzi Orthopedic Institute.
* Cognitively intact
* Inclusion in the rehabilitation program within the Orthopedic Specialist Rehabilitation Unit of IRCCS Galeazzi Orthopedic Institute.
* Informed signed consent.

Exclusion Criteria:

* Cancer history.
* Body Mass Index < 18.5 e > 40.0.
* Melaton consumption.
* Previous clinical sleep disorders.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients undergoing total knee or hip replacement surgery.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Rest-activty Circadian rhythm (RAR) by actigraphy | At baseline untill 10th hospitalization day.
  The 24-hrs daily rhythm of activity levels.
Sleep Efficiency (SE) by actigraphy | At baseline untill 10th hospitalization day.
  The percentage of time in bed spent actually sleeping.
Sleep Latency (SL) by actigraphy | At baseline untill 10th hospitalization day.
  The period of time required for sleep onset after retiring to bed.
Assumed Sleep (AS) by actigraphy | At baseline untill 10th hospitalization day.
  The difference in hours and minutes between the Sleep end and Sleep start times.
Pittsburgh Sleep Quality Index (PSQI) questionnaire | At baseline and at the 10th hospitalization day.
  Evaluation of habitual sleep quality trough a validated questionnaire. 19 items where each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Epworth Sleepiness Scale (ESS) | Every day, from baseline untill the 10th hospitalization day.
  Evaluation of daytime sleepiness. 7 item and each item is weighted on a 0-3 interval scale. Range scores from 0 to 21. Higher scores correspond to higher sleepiness status during the day.

CONTACTS AND LOCATIONS:
Overall Officials: Catia Pelosi, MD, Study Director — IRCCS Galeazzi Orthopedic Institute
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luyster FS, Strollo PJ Jr, Zee PC, Walsh JK; Boards of Directors of the American Academy of Sleep Medicine and the Sleep Research Society. Sleep: a health imperative. Sleep. 2012 Jun 1;35(6):727-34. doi: 10.5665/sleep.1846. PMID 22654183
- [Background] Atkinson G, Davenne D. Relationships between sleep, physical activity and human health. Physiol Behav. 2007 Feb 28;90(2-3):229-35. doi: 10.1016/j.physbeh.2006.09.015. Epub 2006 Oct 25. PMID 17067643
- [Background] de Castro Toledo Guimaraes LH, de Carvalho LB, Yanaguibashi G, do Prado GF. Physically active elderly women sleep more and better than sedentary women. Sleep Med. 2008 Jul;9(5):488-93. doi: 10.1016/j.sleep.2007.06.009. Epub 2007 Aug 30. PMID 17765012
- [Background] Vitale JA, Roveda E, Montaruli A, Galasso L, Weydahl A, Caumo A, Carandente F. Chronotype influences activity circadian rhythm and sleep: differences in sleep quality between weekdays and weekend. Chronobiol Int. 2015 Apr;32(3):405-15. doi: 10.3109/07420528.2014.986273. Epub 2014 Dec 3. PMID 25469597
- [Background] Krenk L, Jennum P, Kehlet H. Sleep disturbances after fast-track hip and knee arthroplasty. Br J Anaesth. 2012 Nov;109(5):769-75. doi: 10.1093/bja/aes252. Epub 2012 Jul 24. PMID 22831887
- [Background] Wylde V, Rooker J, Halliday L, Blom A. Acute postoperative pain at rest after hip and knee arthroplasty: severity, sensory qualities and impact on sleep. Orthop Traumatol Surg Res. 2011 Apr;97(2):139-44. doi: 10.1016/j.otsr.2010.12.003. Epub 2011 Mar 8. PMID 21388906
- [Background] 7. Morin CM, Espie CA. Insomnia: A Clinical Guide to Assessment and Treatment. New York: Springer Science, 2004.
- [Background] Jacobson SA, Dwyer PC, Machan JT, Carskadon MA. Quantitative analysis of rest-activity patterns in elderly postoperative patients with delirium: support for a theory of pathologic wakefulness. J Clin Sleep Med. 2008 Apr 15;4(2):137-42. PMID 18468312